CLINICAL TRIAL: NCT00470821
Title: Randomized, Controlled, Double Blind Trial to Evaluate Sedation and Quality of Life in High-risk, Critically Ill Patients Treated With Oral Melatonin
Brief Title: Oral Melatonin in Critically Ill High-risk Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Giovanni Mistraletti, MD, Istituto di Anestesiologia e Rianimazione, Università di Milano
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Mela-UniMi-0001
Record Dates: First submitted 2007-05-04; First posted 2007-05-08 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-01

CONDITIONS: Critically Ill Patients; Mechanically Ventilated Patients
Keywords: melatonin; actigraphy; sedation; critical patients; ICU
MeSH Terms: interventions — Melatonin; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A - placebo (Placebo Comparator): Identical tablets without the active principles. Each evening, nurses are requested to give 2 tablets at 8 PM and 12 PM
  Interventions: Drug: Placebo
- B - melatonin (Active Comparator): Identical tablets containing melatonin 3 mg Nurses are requested to give two tablets daily, at 8 PM and 12 PM.
  Interventions: Drug: Oral melatonin 3mg BID

INTERVENTIONS:
Drug: Oral melatonin 3mg BID — Identical tablets containing melatonin 3 mg. Nurses are requested to give two tablets daily, at 8 PM and 12 PM
  Other Names: MELATONIN 3 mg
  Arms: B - melatonin
Drug: Placebo — Identical tablets without the active principles. Each evening nurses are requested to give 2 tablets at 8 PM and 12 PM
  Arms: A - placebo

SUMMARY:
Sleep disruptions are extremely common in high-risk critically ill patients. The investigators want to analyse oral melatonin potentialities as a sedative and a free-radicals scavenger for critically ill patients, and secondarily for preventing Delirium during their ICU stay and post-traumatic stress disorders after ICU discharge.

DETAILED DESCRIPTION:
The physiological secretion of such melatonin follows a circadian rhythm: melatonin plasma concentration increases with the dark reaching a peak around to midnight and then gradually decreases (Reiter, 1996; Shigeta et al., 2001; Kunz et al., 2004; Brzezinski et al., 2005).

Administration of oral melatonin could be useful in critically ill high-risk patients in Intensive Care Units because these patients are often suffering from sleep disturbances (Weber et al., 1985; Bourne and Mills, 2004) possibly because of:

* presence of underlying pathology with pain and anxiety,
* presence of oral or nasal respiratory prosthesis,
* execution of therapeutic procedures on 24 h. Moreover it has been demonstrated that in ICU patients melatonin rhythm is desynchronized (Bourne and Mills, 2000). This is probably related to sedation and-or mechanical ventilation. Furthermore, it has been showed that melatonin is a powerful anti-oxidant, therefore it could be potentially useful in critical patients usually characterized by increased production of oxygen free radicals.

AIM OF THE STUDY The study is aimed to estimate if the administration of oral melatonin in ICU patients is able to regularize the sleep-waking rhythm, improving sleep quality and reducing episodes of agitation/mental confusion. The main objectives are: assessment of sleep quality, prevalence of mental confusion/agitation, amount of daily sedative drugs administered and modification of redox status.

ENROLLMENT OF PATIENTS At the admission in ICU, obtained the informed consent, the patients will be randomly assigned to the "Treatment" group receiving melatonin 3mg BID by oral route (or nasogastric tube) or to the "Control" group receiving placebo. The sedation will be performed according to clinical standard.

EXPERIMENTAL PROTOCOLS

The following parameters will be monitored:

* epidemiological data,
* quality of the sleep estimated by wrist actigraphy,
* EEG profile on 24h in order to estimate the distribution of sleep phases,
* diurnal and nocturnal hours of sleep,
* total amount of sedative drugs during 24 hours, particularly during nocturnal sedation,
* assessment of sedation level (RASS) (Sessler et al., 2002; Ely et al., 2003),
* episodes of psychomotor agitation and mental confusion (CAM-ICU) (Ely, 2001; 2004),
* evaluation of blood redox state (GSH, GSSG, GSH/GSSG),
* adverse events.

AT THE DISCHARGE FROM ICU, evaluation of:

* SCID-I and SCID-II (Structured Clinical Interview for DSM),
* CAPS (Clinician Administered PTSD Scales),
* HAM-A and HAM-D (Hamilton Rating Scales for Anxiety and for Depression),
* completion of the module for the stressors in ICU and for the transcription of the dreams.

  3 MONTHS AFTER DISCHARGE FROM ICU, evaluation of:
* SCID-I and II,
* CAPS,
* HAM-A and HAM-D,
* TAT (Thematic Apperception Test),
* completion of the module for the stressors in ICU and for the transcription of the dreams.

ELIGIBILITY:
Inclusion Criteria:

* High Treatment > 1 day
* Normal gastrointestinal function

Exclusion Criteria:

* Status asthmaticus
* Chronic renal failure under dialytic treatment
* Severe hepatopathy (Child-Pugh class = C)
* Comatous patients (GCS < 12)
* Head trauma, severe neurological diseases (ictus cerebri, SAH, ...)
* Intoxicated patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2007-05; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Overall sedatives daily doses | Discharge from ICU

SECONDARY OUTCOMES:
Prevalence of Delirium assessed with CAM-ICU | Discharge from ICU
Prevalence of mental disorders | 60 days after ICU discharge
ICU length of stay | Discharge from ICU
ICU mortality | Discharge from ICU
Hospital mortality | Hospital discharge
Sleep quantity assessed by wrist actigraphy | Discharge from ICU

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Iapichino, MD, Study Chair — University of Milan
Locations (1):
- Azienda Ospedaliera San Paolo - Polo Universitario, Milan, Italy